CLINICAL TRIAL: NCT06927960
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Dose Escalation Study in Subjects to Evaluate the Safety, Tolerability and Pharmacokinetics of AH-001 Following Topical Single and Multiple Ascending Dose Administration
Brief Title: Evaluation of the Safety, Tolerability and Pharmacokinetics of AH-001 Following Topical Single and Multiple Ascending Dose Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AnHorn Medicines Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AH-001-01
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia | interventions — AH 001

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 2% AH-001 (Experimental)
  Interventions: Drug: AH-001 or placebo
- 1% AH-001 (Experimental)
  Interventions: Drug: AH-001 or placebo
- 0.5% AH-001 (Experimental)
  Interventions: Drug: AH-001 or placebo
- 0.2% AH-001 (Experimental)
  Interventions: Drug: AH-001 or placebo

INTERVENTIONS:
Drug: AH-001 or placebo — SAD: Subjects are planned to receive a single dose of AH-001 or placebo once MAD: Subjects are planned to receive a single daily dose of AH-001 or placebo for 7 consecutive days

SUMMARY:
The goal of this clinical trial is to assess the safety of the AH-001 drug substance at concentrations of 0.2%, 0.5%, 1%, and 2% in healthy volunteers and male subjects with androgenetic alopecia (AGA).

Primary objective:

* To evaluate the safety, tolerability, and pharmacokinetics profiles of a single ascending dose (SAD) of AH-001 in healthy volunteers.
* To evaluate the safety, tolerability, and pharmacokinetics profiles of multiple ascending doses (MAD) of AH-001 in male subjects with androgenetic alopecia (AGA).

ELIGIBILITY:
Inclusion Criteria at Screening

Subjects must meet the following criteria to be eligible for participation in the study:

For all (Cohort 1~8):

1. Age range: 18 to 65 years.
2. Body weight: ≥ 50 kg for males, ≥ 45 kg for females; Body Mass Index (BMI) 19 to 30 kg/m2 (inclusive).
3. Subjects understand and agree to comply with planned study procedures, can communicate well with the investigator, understand the requirements of the study, and have provided written informed consent.
4. Following the assessment, the principal investigator considered the individual healthy, including a detailed medical history, complete physical examination, clinical laboratory tests, 12-lead ECG, and vital signs evaluation.
5. No history of excessive sensitivity or allergic reactions to topical formulations.

For Cohort 1~4 (SAD):

1. Healthy subjects, including males or non-pregnant, non-breastfeeding females.
2. The skin of the upper arm must be healthy without damage or wound.
3. Treatment sites (upper arm skin) must be free of scars, tattoos, or dermatological defects that might impair measurements.

For Cohort 5~8 (MAD):

1. Male subjects with a clinical diagnosis of mild to severe AGA; rating III to VII (contains III Vertex, IIIa, IVa, and Va) on the modified Norwood Hamilton Scale, with a history of ongoing hair loss.
2. Willingness to maintain the same hairstyle, hair length, hair color, and hair care regimen throughout the study.
3. The skin of the scalp must be healthy without damage or wounds.
4. Treatment sites (scalp skin) must be free of scars, tattoos, or dermatological defects that might impair measurements.

Exclusion Criteria at Screening

Subjects are excluded from this study if any 1 or more of the following criteria is met:

For all (Cohort 1~8):

1. History of allergy to the investigational drug or its components.
2. Individuals who used systemic treatment (including finasteride, oral minoxidil, dutasteride or similar products) that is known to or reasonably believed in the opinion of the Investigator to affect hair growth within the last 3 months prior to dosing.
3. Presence of any visible skin disease, damage, or condition at the application site that, in the investigator's opinion, may jeopardize subject safety or interfere with the assessment of the test site reaction.
4. Clinical history of clinically significant disorders in various systems (including gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, and lipid metabolism) that may limit the ability to assess the associated adverse events based on Investigational judgement or known or suspected malignancy.
5. Positive blood screen for human immunodeficiency virus (HIV) or syphilis. Positive blood screen for active infection of hepatitis B or hepatitis C
6. Hospital admission or planned or anticipated major surgical procedure that would interfere with the ability to comply with protocol requirement within 30 days prior to screening.
7. Participation in another investigational drug trial within 3 months before the first dosing.
8. History of prescription drug abuse or illicit drug use within 6 months prior to screening or a positive screen for drugs of abuse.
9. Excessive alcohol consumption (>14 units per week, 1 unit of alcohol ≈ 360 mL of beer or 45 mL of spirits containing 40% alcohol or 150 mL of wine) within 3 months prior to signing the informed consent form, or a positive breath or urine alcohol test results the day before dosing, or inability to abstain from alcohol during the study.
10. Chronic consumption of excessive tea, coffee, or caffeine-containing beverages (>8 cups per day, 1 cup = 240 mL) within 6 months before dosing.
11. Consumption of caffeine, alcohol, xanthine, or grapefruit-containing beverages within 48 hours the first dose and stay-on-site period.
12. Difficulty with blood collection, intolerance to venipuncture, or a history of needle phobia or hemophobia.
13. Blood donation from 7 days before the first dosing until 2 days after the last dosing. Loss of ≥450 mL of blood within 3 months before the first dosing.
14. Smoking more than 5 cigarettes per day within 3 months before the study and inability to stop smoking within 7 days before the first dosing until 2 days after the last dosing.
15. Use of prescription or over-the-counter medications and herbal supplements (including St John's Wort, herbal teas, and garlic extracts) within 30 days before the first dosing until 2 days after the last dosing (except for paracetamol/acetaminophen, ibuprofen, and hormonal contraceptives).
16. For females of childbearing potential: Unwillingness to use a highly effective contraceptive method (method of birth control which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, non-hormonal or hormonal intrauterine devices (IUDs), sexual abstinence or vasectomized partner) during sexual intercourse with a partner of childbearing potential throughout the study and for 1 month after its completion. Only males capable of reproduction are required to use a reliable form of contraception throughout the study and for 1 month after study completion (vasectomized males of at least 6 months are exempt).
17. Employment or affiliation with the investigator, study site, sponsor, or contract research organization.
18. Other conditions affecting compliance, as determined by the investigator, or inability to participate in the study for personal reasons.
19. Inability to communicate or cooperate with healthcare professionals due to neurological, psychiatric, or language disorders.

For Cohort 5~8 (MAD):

1. Subjects with dermatological disorders of the scalp in the target region that may interfere with the application of the investigational drug-such as fungal or bacterial infections, seborrheic dermatitis, psoriasis, eczema, folliculitis, scars, or scalp atrophy-or with skin pathology or conditions that could affect the evaluation of the investigational drug or require interfering therapy, including topical, systemic, or surgical treatments.
2. Genetic disorders affecting hair growth or patterns or requiring certain treatments.
3. History of hair weaves, non-breathable wigs, hair transplant or hair bonding that will interfere with applying the investigational drug or observing safety and tolerability.
4. History of active hair loss due to conditions other than AGA, such as diffuse telogen effluvium, alopecia areata, scarring alopecia, or trichotillomania.
5. Severe dietary or weight changes within the past six months, or a history of eating disorders that has contributed to hair loss in the opinion of the Investigator.
6. Subjects that used topical scalp treatments for the management of hair loss (including minoxidil, anti-androgens) or a history of radiation of the scalp within the last 4 weeks prior to dosing.
7. Unstable disorders in various systems that could affect subject safety throughout the study, as determined by the investigator.

Exclusion Criteria at Admission

Subjects will not be administered with study drug if they meet any of the following rules at admission:

1. Any abnormal laboratory values at admission: Hb <12.0g/dL for women and < 13.0 g/dL for men, WBC < 3,000 cells/mm3, absolute neutrophil count < 1,500 cells/mm3, platelet count < 100,000 cells/mm3, serum creatinine ≥ 2 mg/dL, ALT or AST levels ≥ 2 x ULN, total bilirubin ≥ 1.5 x ULN, Prothrombin Time (PT) ≥ 1.5 x ULN
2. Any abnormal laboratory values that are considered clinically significant by the Investigator at admission
3. Any clinically significant abnormality on 12-lead ECG or a QT interval corrected with the Fridericia formula (QTcF) greater than 450 msec for females and 430 msec for males at admission
4. Positive urine drug screen or breath test at admission
5. If female, positive serum pregnancy test at admission
6. Acute illness within 2 weeks before dosing, unless approved by the Sponsor's Medical Monitor

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2025-03-24 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Number and percentage of subjects with treatment-emergent adverse events | From the first dose until 2 days after the last dose
Changes from baseline in local skin reaction | From the first dose until 2 days after the last dose
Pharmacokinetic characterization of Cmax for AH-001 | From the first dose until 2 days after the last dose
Pharmacokinetic characterization of Tmax for AH-001 | From the first dose until 2 days after the last dose
Pharmacokinetic characterization of AUC for AH-001 | From the first dose until 2 days after the last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences Clinical Los Angeles, Inc., Los Angeles, California, United States